CLINICAL TRIAL: NCT00241631
Title: Enhancement of In-vitro GC Function in Patients With COPD. A Randomised, Double Blind, Placebo Controlled, Parallel-group Study to Investigate the Effect of Theophylline and Fluticasone on Induced Sputum Cells Obtained Form COPD Patients
Brief Title: Enhancement of in-Vitro GC Function in Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Tanabe Pharma Corporation (Industry); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mitHDAC#1
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Theophylline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Inhaled Theophylline placebo capsule, then placebo, then active Theophylline
  Interventions: Drug: placebo; Drug: Theophylline
- Steroid (Active Comparator): Inhaled Theophylline placebo capsule, then Fluticasone Propionate 500 ug bid, then active Theophylline
  Interventions: Drug: Fluticasone Propionate; Drug: Theophylline

INTERVENTIONS:
Drug: Fluticasone Propionate — 500 u
  Arms: Steroid
Drug: placebo
  Arms: Placebo
Drug: Theophylline — Theophylline placebo capcule

SUMMARY:
The investigator wish therefore to continue these studies on theophylline principally by conducting a small clinical pilot study on 20-30 COPD patients in a randomised, double-blind, placebo-controlled, parallel-group study.

DETAILED DESCRIPTION:
The global burden of COPD - a common and debilitating chronic inflammatory disease that is characterised by the progressive development of airflow limitation (shortness of breath - SOB) and is poorly reversible with currently available drugs -is increasing. Cigarette smoking is strongly linked with the ongoing inflammation; inflammation that can continue even when the patient has stopped smoking. The severity of airflow limitation (SOB) is correlated with the degree of pulmonary (lung) inflammation.

Histone deacetylases (HDACs)are important molecules in suppressing this pulmonary inflammation. We have recently shown that patients with COPD have a reduction in total HDAC which correlates with the severity of their lung disease.

Corticosteroids (anti-inflammatory treatment) act, at least in part, by recruitment of these HDACs to the site of active inflammatory gene transcription (which reduces the production of inflammatory molecules) and are widely used in COPD in patients with severe disease. Unfortunately, in COPD, inhaled corticosteroids seem to have little effect on the underlying inflammation (though in a selective group of patients with COPD they do reduce the number of infections a patient may have by a small amount).

Theophylline has been used in the treatment of asthma and COPD for over 70 years, but its use has recently declined. Data so far obtained in primary cells (cells from patients used in the laboratory) from COPD patients suggests that low dose theophylline (~5mg/l) should be effective in restoring steroid sensitivity in patients with COPD (and hence reduce inflammation thus improving SOB).

ELIGIBILITY:
Inclusion Criteria:Participants with COPD with an FEV1 of 80-30% predicted. This will incorporate the majority of participants with COPD seen within the chest clinic. Patients with an FEV1 > 80% predicted are not generally severe enough to warrant hospital follow up. These patients are also unlikely to have severe enough disease (and therefore airway inflammation) which may be modified by the therapeutic agents we are studying.

Patients with an FEV1 < 30% tend to have more severe symptom limitation and generally (though not always) find participation in a clinical trial involving 4 visits to the clinic difficult. Their airway disease is also generally less responsive to therapeutic intervention and as a consequence finding measurements which show changes to these therapeutic interventions is more difficult.

COPD patients

* All participants will be classified to Stage 2-3 of the GOLD (Global initiative for Obstructive Lung Disease) guidelines
* Male or female, aged 45-80 years (according to GOLD guidelines)
* 30% < FEV1 < 80% predicted
* FEV1/FVC < 70%
* Cigarette exposure of >10 pack-years#
* With or without chronic symptoms (cough, sputum production, dyspnea).
* Steroid therapy will be stopped before run-in, but long acting bronchodilators are acceptable.
* The participants are able to give informed consent # The smoking history should include both the number smoked, for how long, and an estimate of total pack-years of smoking. One pack of 20 cigarettes smoked per day for 1 year = one pack year. Total pack years = No. cigarettes smoked per day/20 x no. years of smoking

Exclusion Criteria:

Any history or evidence of asthma

* Pregnancy, breast-feeding or planned pregnancy during the study. Fertile women not using acceptable contraceptive measures, as judged by the investigator
* Hospital admission with respiratory infection within the last 6 months
* Upper respiratory infection within the last 4 weeks
* Participants who have received research medication within the previous one month
* Participants unable to give informed consent
* Any mental condition rendering the participant unable to understand the nature, scope and possible consequences of the study
* Known or suspected hypersensitivity to study therapy or excipients
* Participants with significant or unstable ischemic heart disease, arrhythmia, cardiomyopathy, heart failure, uncontrolled hypertension as defined by the investigator, or any other relevant cardiovascular disorder as judged by the investigator
* Any current respiratory tract disorders other than COPD, which is considered by the investigator to be clinically significant
* Any significant disease or disorder (e.g. gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) or abnormality laboratory tests which, in the opinion of the investigator, may either put the participant at risk because of inclusion in the study, or may influence the results of the study, or the participants ability to take part in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ian adcock, PhD, Principal Investigator — Imperial College London
Locations (1):
- Windsor chest clinic KEVII Hospital, Windsor, Berks, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ito K, Ito M, Elliott WM, Cosio B, Caramori G, Kon OM, Barczyk A, Hayashi S, Adcock IM, Hogg JC, Barnes PJ. Decreased histone deacetylase activity in chronic obstructive pulmonary disease. N Engl J Med. 2005 May 12;352(19):1967-76. doi: 10.1056/NEJMoa041892. PMID 15888697
- [Result] Ford PA, Durham AL, Russell RE, Gordon F, Adcock IM, Barnes PJ. Treatment effects of low-dose theophylline combined with an inhaled corticosteroid in COPD. Chest. 2010 Jun;137(6):1338-44. doi: 10.1378/chest.09-2363. Epub 2010 Mar 18. PMID 20299628
- [Derived] Kirkham PA, Whiteman M, Winyard PG, Caramori G, Gordon F, Ford PA, Barnes PJ, Adcock IM, Chung KF. Impact of theophylline/corticosteroid combination therapy on sputum hydrogen sulfide levels in patients with COPD. Eur Respir J. 2014 May;43(5):1504-6. doi: 10.1183/09031936.00131513. Epub 2014 Feb 13. No abstract available. PMID 24525446

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Inhaled Theophylline placebo capsule, then inhaled placebo, then active Theophylline
Period: Run in (2 Weeks)
Arm/Group | Placebo | Steroid
Started | 25 | 24
Completed | 22 | 21
Not Completed | 3 | 3
Not completed — Physician Decision | 3 | 3
Period: Phase 1 (4 Weeks)
Arm/Group | Placebo | Steroid
Started | 22 | 21
Completed | 14 | 16
Not Completed | 8 | 5
Not completed — sore throat | 1 | 0
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Lack of Efficacy | 0 | 1
Period: Wash Out (2 Weeks)
Arm/Group | Placebo | Steroid
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0
Period: Phase 2 (4 Weeks)
Arm/Group | Placebo | Steroid
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Steroid | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (2.2) | 69 (1.9) | 65 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 11 | 14 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Sputum Inflammatory Cell Counts
Description: Supernatant collect, cell pellets count on slides
Time Frame: 10 weeks
Population: Using marginal means as results
Measure: Mean (95% Confidence Interval); unit: millions cells/ ml
Arm/Group | Placebo | Steroid
Number analyzed (Participants) | 14 | 16
millions cells/ ml | 5.42 [3.56 to 8.2] | 3.89 [2.6 to 5.76]
Statistical Analysis 1: Comparison: Placebo vs Steroid; Test type: Superiority; p = 0.012, Mixed Models Analysis

2. Secondary Outcome: Interleukin 8 (IL8)
Description: Interleukin 8 (IL8) assessed from sputum
Time Frame: 10 weeks
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Placebo | Steroid
Number analyzed (Participants) | 14 | 16
ng/mL | 33.3 [20 to 56] | 28.3 [19 to 42]
Statistical Analysis 1: Comparison: Placebo vs Steroid; Test type: Superiority; p < 0.05, Mixed Models Analysis — calculated

3. Secondary Outcome: Total Sputum Eosinophils
Description: Total eosinophils cells assessed from sputum
Time Frame: 10 weeks
Measure: Mean (95% Confidence Interval); unit: millions cells/ml
Arm/Group | Placebo | Steroid
Number analyzed (Participants) | 14 | 16
millions cells/ml | 0.132 [0.09 to 0.2] | 0.053 [0.03 to 0.1]
Statistical Analysis 1: Comparison: Placebo vs Steroid; Test type: Superiority; p < 0.05, Mixed Models Analysis — calculated

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Placebo | Steroid
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Steroid (N=16)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) — Nausea and upset stomach

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes